CLINICAL TRIAL: NCT01554891
Title: Reliability and Initial Validation of the INTRuST Structured Assessment For Evaluation of TBI (SAFE-TBI)
Brief Title: INTRuST Structured Assessment For Evaluation of TBI (SAFE-TBI)
Acronym: SAFE-TBI
Status: Completed | Type: Observational
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: INTRuST-SAFE-TBI
Record Dates: First submitted 2012-03-12; First posted 2012-03-15 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Brain Injuries, Traumatic
Keywords: brain injuries, traumatic; military personnel; classification; diagnosis; instrumentation
MeSH Terms: conditions — Brain Injuries, Traumatic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cohort 1: 100 OEF/OIF/OND veterans returning to Joint Base Lewis-McChord and Fort Bragg who screen positive for TBI on the Post Deployment Health Assessment (PDHA) TBI screen
- Cohort 2: 100 OEF/OIF/OND veterans seeking care at Northern New England VA Research Consortium (NNEVARC) VA Medical Centers (VAMCs) who screen positive for TBI on VA Level 1 TBI screen
- Cohort 3: 200 participants in WRNMMC and Fort Belvoir Community Hospital Brain Indices Study (100 with mild TBI; 100 without mild TBI).

SUMMARY:
The current study will evaluate the initial reliability and validity of a new instrument, the INTRuST Structured Assessment for Evaluation of TBI (SAFE-TBI), in three samples of Operation Enduring Freedom/Operation Iraqi Freedom/Operation New Dawn (OEF/OIF/OND) veterans. The SAFE-TBI is a relatively brief measure developed by INTRuST consortium investigators and designed to be given by a trained administrator. It allows for a determination of the level of evidence for exposure to a mild traumatic brain injury (TBI) using the following categories: Strong, Moderate, Weak, or No Evidence of mild TBI. The first objective is to determine the reliability (both test-retest and inter-rater) in a sample of 100 veterans recently returned from deployment at Joint Base Lewis-McChord and Fort Bragg (Cohort 1), who have screened positive for TBI on the Post-Deployment Health Assessment. The second objective is to determine the concordance between the SAFE-TBI and the VA TBI Screen in 100 OEF/OIF/OND veterans within the Northern New England VA Research Consortium (Cohort 2). The third objective, to be carried out in a sample of 200 Walter Reed National Military Medical Center (WRNMMC) and Fort Belvoir Community Hospital OEF/OIF/OND patients (Cohort 3), is to determine the sensitivity and specificity of the SAFE-TBI using the INTRuST study "Brain Indices of Risk for Posttraumatic Stress Disorder after Mild Traumatic Brain Injury" initial evaluation as the "gold standard" for TBI assessment.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

1. Military personnel returning to Joint Base Lewis-McChord and Fort Bragg from deployment in support of OEF/OIF/OND between the ages of 18-60.
2. Screen positive on the PDHA TBI screen and referred to the Madigan Army Medical Center TBI clinic and Womack Army Medical Center.
3. Capable of giving informed consent.

Cohort 2:

1. Veterans of OEF/OIF/OND between the ages of 18-60, receiving care at any of the three VAMCs that comprise the Northern New England VA Research Consortium (White River Junction, VT; Manchester, NH; Togus, ME).
2. Screen positive on the VA Level 1 TBI screen.
3. Capable of giving informed consent.

Cohort 3:

Military Personnel participating in the INTRuST Consortium Brain Indices Study at Walter Reed National Military Medical Center and Fort Belvoir Community Hospital. This study has the following Inclusion Criteria:

1. Must be a patient at WRNMMC or FBCH
2. Must be Defense Enrollment Eligibility Reporting System (DEERS) eligible.
3. Must be diagnosed TBI positive or certified as TBI negative by a licensed medical practitioner using Department of Defense (DoD) criteria
4. For mTBI subjects, an initial score of 13-15 on the Glasgow Coma Scale
5. Aged 18-60

Exclusion Criteria:

Cohort 1:

1. Speech/language deficit of sufficient severity to preclude answering interview questions
2. Unable or unwilling to provide informed consent and Health Insurance Portability and Accountability Act (HIPAA)authorization ("unable" includes cases in which the potential subject cannot read and understand English well enough to provide informed consent).

Cohort 2:

1. Speech/language deficit of sufficient severity to preclude answering interview questions.
2. Unable or unwilling to provide informed consent and HIPAA authorization ("unable" includes cases in which the potential subject cannot read and understand English well enough to provide informed consent).
3. Second level in-depth TBI evaluation done prior to SAFE TBI interview

Cohort 3:

Exclusion criteria for Cohort will be those used in the WRNMMC and Fort Belvoir Community Hospital Brain Indices Study as follows:

1. Unable or unwilling to provide informed consent and HIPAA authorization ("unable" includes cases in which the potential subject cannot read and understand English well enough to provide informed consent).
2. Penetrating head injury.
3. Record of drug or alcohol abuse or dependence in the past six months as documented in medical chart.
4. Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders -IV (SCID) reveals current or lifetime PTSD diagnosis related to life events that occurred prior to most recent deployment.
5. Taking intravenous medications for pain; participation will be delayed until such medication has been discontinued.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cohort 1: Active duty OEF/OIF/OND military personnel ages 18-60 who have recently screened positive for TBI following deployment.
  Cohort 2: OEF/OIF/OND veterans ages 18-60 who have recently screened positive for TBI.
  Cohort 3: Participants ages 18-60 in the INTRuST Consortium Brain Indices Study at WRNMMC or FBCH.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2012-02; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Flashman, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (6):
- United States (6):
  - Walter Reed National Military Medical Center, Washington D.C., District of Columbia
  - Togus VA Medical Center, Augusta, Maine
  - Manchester VA Medical Center, Manchester, New Hampshire
  - White River Junction VA Medical Center, White River Junction, Vermont
  - Fort Belvoir Community Hopsital (FBCH), Fort Belvoir, Virginia
  - Madigan Army Medical Center, Fort Lewis, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This difference is due to screened patients who were enrolled, but then found ineligible,were unreachable, or withdrew from study.
Groups:
- Test-Retest Reliability of SAFE-TBI: 100 OEF/OIF/OND veterans returning to Joint Base Lewis-McChord and Fort Bragg who screen positive for TBI on the Post Deployment Health Assessment (PDHA) TBI screen.
  This component of the project assessed test-retest reliability (4-6 weeks), as well as the eﬀects of diﬀerent raters; Research Coordinators (TRCs) vs. experienced TBI Clinicians (TBICs) at the Madigan Army Medical Center (MAMC) TBI Clinic. Cohort 1 included subjects recently returned from deployment in Iraq or Afghanistan to Joint Base Lewis-McChord or veterans served at the White River Junction and Togus VAMC who screened positive for TBI on the PDHA. After the initial interview, the SAFE-TBI will be administered for the second time 4-6 weeks later. Participants were assigned to one of four assessment paradigms (i. TRC time 1 and TBIC time 2; ii. TRC time 1 and TRC time 2; iii. TBIC time 1 and TBIC time 2; or iv. TBIC time 1 and TRC time 2).
- Comparison of SAFE-TBI and VA Screen: 100 OEF/OIF/OND veterans seeking care at Northern New England VA Research Consortium (NNEVARC) VA Medical Centers (VAMCs) who screen positive for TBI on VA Level 1 TBI screen This component of the project assessed the correlation of the VA TBI Level 1 screen with the SAFE-TBI.
  Participants were OEF/OIF/OND veterans (seeking care at the Northern New England VA Research Consortium [NNEVARC]) that screen positive for TBI on the VA screen when seeking treatment at the VA. Prior to the second level in-depth TBI evaluation, they were interviewed by a TRC using SAFE-TBI.
- Sensitivity and Specificity of SAFE-TBI: 200 participants in WRNMMC and Fort Belvoir Community Hospital Brain Indices Study (100 with mild TBI; 100 without mild TBI).
Period: Overall Study
Arm/Group | Test-Retest Reliability of SAFE-TBI | Comparison of SAFE-TBI and VA Screen | Sensitivity and Specificity of SAFE-TBI
Started | 105 | 120 | 57
Completed | 98 | 115 | 55
Not Completed | 7 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Test-Retest Reliability of SAFE-TBI: 100 OEF/OIF/OND veterans returning to Joint Base Lewis-McChord and Fort Bragg who screen positive for TBI on the Post Deployment Health Assessment (PDHA) TBI screen
- Comparison of SAFE-TBI and VA Screen: 100 OEF/OIF/OND veterans seeking care at Northern New England VA Research Consortium (NNEVARC) VA Medical Centers (VAMCs) who screen positive for TBI on VA Level 1 TBI screen
- Total: Total of all reporting groups
Arm/Group | Test-Retest Reliability of SAFE-TBI | Comparison of SAFE-TBI and VA Screen | Sensitivity and Specificity of SAFE-TBI | Total
Number analyzed (Participants) | 98 | 115 | 55 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.29 (9.30) | 33.03 (8.68) | 29.20 (8.56) | 31.33 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 19
  Male | 91 | 109 | 49 | 249
Presence of TBI [Number; unit: participants] — Cohort 1: the degree of agreement for SAFE-TBI outcome (no evidence of TBI vs. at least, weak evidence of TBI) across the two assessment time points (initial vs. 4 to 6 weeks), as well as the two rater types TRC vs. TBIC Cohort 2:the distribution of SAFE-TBI outcome (percent assigned to each evidence category of the SAFE-TBI) in a group of veterans who have screened positive on the VA TBI screen.
  Cohort 3:Gold Standard comparison; the sensitivity and speciﬁcity of the SAFE-TBI to identify individuals with TBI
  participants | 91 | 115 | 55 | 261

OUTCOME MEASURES:

1. Primary Outcome: Test-retest Reliability SAFE-TBI
Description: Reliability of SAFE-TBI, as determined by test-retest and inter-rater reliability, in a sample of 100 veterans recently returned from deployment (Cohort 1) Cohort 1: The primary endpoints for this sub-study (cohort) are the degree of agreement for SAFE-TBI outcome (no evidence of TBI vs. at least, weak evidence of TBI) across the two assessment time points (initial vs. 4 to 6 weeks) as well as the two rater types TRC vs. TBIC. (Speciﬁc Aim 1).
Time Frame: Up to 6 weeks
Population: Analyses done on Cohort 1, and a subset of Cohort 2 and 3 who got repeat interview.
Measure: Number (95% Confidence Interval); unit: kappa (reliability)
Groups:
- Test-Retest Reliability of SAFE-TBI: Cohort 1 was used to determine test-retest reliability of the SAFE-TBI instrument.
Arm/Group | Test-Retest Reliability of SAFE-TBI
Number analyzed (Participants) | 98
kappa (reliability)
  Cutoff 1 (no vs. at least weak evidence) | 0.372 [0.055 to 0.69]
  Cutoff 2 (no or weak vs. at least moderate evid) | 0.504 [0.298 to 0.711]
  Cutoff (no, weak, moderate vs. strong) | 0.581 [0.412 to 0.75]

2. Primary Outcome: Concordance Rate of Current VA Screening Instruments and the SAFE-TBI.
Description: Concordance rate of current VA TBI screening instruments and the SAFE-TBI in 100 OEF/OIF/OND veterans who have screened positive for TBI (Cohort 2) Cohort 2: The primary endpoint for this sub-study is the distribution of SAFE-TBI outcome (percent assigned to each evidence category of the SAFE-TBI) in a group of veterans who have screened positive on the VA TBI screen. (Speciﬁc Aim 2).
Time Frame: baseline
Population: Analyses done for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Comparison of SAFE-TBI and VA Screen: Veterans
Arm/Group | Comparison of SAFE-TBI and VA Screen
Number analyzed (Participants) | 115
percentage of participants
  Strong Evidence | 64.35 [55.59 to 73.1]
  Moderate Evidence | 11.3 [5.52 to 17.09]
  Weak Evidence | 14.78 [8.3 to 21.27]
  No Evidence | 9.57 [4.19 to 14.94]

3. Primary Outcome: Sensitivity and Specificity of the SAFE-TBI
Description: Sensitivity = True Positives/(True Positive + False Negatives) Specificity = True Negatives/(True Negative + False Positives) Cutoff 2 = At least moderate evidence of TBI vs. no or weak evidence of TBI
Time Frame: 6-months after medical evacuation
Population: Data were only collected for cohort 3.
Measure: Number; unit: percentage
Groups:
- Sensitivity and Specificity of SAFE-TBI: Sensitivity = True Positives/(True Positive + False Negatives) Specificity = True Negatives/(True Negative + False Positives)
Arm/Group | Sensitivity and Specificity of SAFE-TBI
Number analyzed (Participants) | 55
percentage
  Sensitivity for Cutoff 2 | 93
  Specificity for Cutoff 2 | 50

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Test-Retest Reliability of SAFE-TBI | Comparison of SAFE-TBI and VA Screen | Sensitivity and Specificity of SAFE-TBI
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/115 | 0/55
Other Adverse Events (participants affected / at risk) | 0/98 | 0/115 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No